CLINICAL TRIAL: NCT01544465
Title: Effect of a Structured Physical Activity Program on Sleep Quality and Sleepiness in Parkinson's Disease
Brief Title: Structured Physical Activity for Sleep Quality and Daytime Sleepiness in Patients With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting, funding lapsed
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Roneil Malkani, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00045490; 67-PA-11 (Other Grant/Funding Number: American Sleep Medicine Foundation)
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease; Poor Quality Sleep; Hypersomnia
Keywords: Parkinson's disease; Sleep Quality; Daytime sleepiness; physical therapy; exercise
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured physical activity (Experimental): Rehabilitation evaluation followed by physical therapy for approximately 8 weeks
  Interventions: Behavioral: Structured Physical Activity
- Sleep hygiene education (Active Comparator): Sleep hygiene education consists of educational materials on insomnia published by the American Academy of Sleep Medicine.
  Interventions: Behavioral: Structured Physical Activity; Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Structured Physical Activity — Rehabilitation evaluation and 8 weeks of physical therapy
Behavioral: Sleep hygiene education — Educational materials on insomnia published by the American Academy of Sleep medicine
  Other Names: Review of sleep hygiene checklist every 2 weeks via telephone for 8 weeks.
  Arms: Sleep hygiene education

SUMMARY:
The purpose of this study is to examine the ability of a structured physical activity program to improve sleep quality and daytime sleepiness in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic, progressive, neurodegenerative disease that affects 1% of elderly people. Sleep disturbances affect up to 88% of patients with PD and commonly include sleep fragmentation and excessive daytime sleepiness (EDS); these symptoms can significantly impair quality of life. The cause of sleep fragmentation and EDS is likely multifactorial, including medications, neurodegeneration, primary sleep disorders such as sleep apnea, and decreased physical activity. Pharmacotherapy in this population is limited due to side effects and drug-drug interactions.

The goal of this project is to develop non-pharmacologic therapies for impaired sleep quality and EDS in PD. Sleep disturbances and EDS are common among patients with PD and negatively affect their quality of life. There is data to support a role for physical activity in sleep in older adults with and without insomnia. Additionally, increased physical activity in patients with PD has been associated with improvement in PD motor symptoms and quality of life. Therefore, the investigators propose to examine the ability of structured physical activity to improve sleep quality and daytime sleepiness in patients with PD.

The overall objective of the proposed project is to develop behavioral approaches to improve sleep quality and daytime function in PD. The investigators propose to examine the effect of a structured physical activity program and sleep hygiene education on nighttime sleep quality and EDS in patients with idiopathic PD. There will be two groups: 1) a structured physical activity program with sleep hygiene education (SPA group), and 2) a control group receiving only sleep hygiene education (SH group) who will be offered the delayed physical activity program.

The investigators hypothesize that the structured physical activity program will improve subjective and objective sleep quality and daytime sleepiness compared to sleep hygiene education alone.

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of Hoehn and Yahr stage I to III idiopathic Parkinson's disease,
* Male and female.
* Age of onset of PD >= 50 years;
* Impaired sleep quality determined by Parkinson's disease sleep scale (PDSS-2) total score ≥ 12;
* EDS as determined by Epworth Sleepiness Scale (ESS) > 10;
* Sedentary (< 30 minutes/day or < 2 times/week of exercise) based on physical activity history;
* Stable on medications for PD for at least 2 months;
* After clinical evaluation, was provided with a referral by their Movement Disorders Neurologist for an evaluation at the Movement Disorders Rehabilitation Evaluation Clinic at the Rehabilitation Institute of Chicago.

Exclusion Criteria:

* Cognitive impairment as determined by Montreal Cognitive Assessment (MoCA) total score < 25;
* High likelihood of sleep disordered breathing as determined by the Berlin Questionnaire (BQ);
* Restless legs syndrome (RLS) based on the International RLS Study Group diagnostic criteria;
* Current use of any sedative/hypnotics or stimulants, tricyclic antidepressants, and trazodone;
* Use of selective serotonin reuptake inhibitors (SSRIs) and bupropion will be allowed only if the patient has been on a stable dose for at least three months;
* Unstable medical or psychiatric condition;
* History of falls in the last 2 months;
* Participants with parasomnias such as Rapid Eye Movement Behavior Disorder will not be excluded as up to 50% of patients with PD have parasomnias and exclusion of these patients would result in difficulty with recruitment and the results would be less generalizable;
* Current depression based on BDI-II total score > 19;
* Current occupation involves shift work;
* At visit #2, Apnea-hypopnea index >15 on baseline PSG;
* At visit #2, Periodic limb movements in sleep index >15 on baseline PSG;
* At physiatry evaluation at RIC, inpatient rehabilitation is recommended.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in polysomnographically-derived wake after sleep onset | Baseline and 10 weeks
Change in mean sleep latency test-derived mean sleep latency | Baseline and 10 weeks

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index | Baseline and 10 weeks
  The Pittsburgh Sleep Quality Index is a survey-derived measure of sleep quality.
Change in Epworth Sleepiness Scale | Baseline and 10 weeks
  The Epworth Sleepiness Scale is a survey-derived measure of sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis C Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Hirtz D, Thurman DJ, Gwinn-Hardy K, Mohamed M, Chaudhuri AR, Zalutsky R. How common are the "common" neurologic disorders? Neurology. 2007 Jan 30;68(5):326-37. doi: 10.1212/01.wnl.0000252807.38124.a3. PMID 17261678
- [Background] Menza M, Dobkin RD, Marin H, Bienfait K. Sleep disturbances in Parkinson's disease. Mov Disord. 2010;25 Suppl 1(Suppl 1):S117-22. doi: 10.1002/mds.22788. PMID 20187236
- [Background] Ondo WG, Dat Vuong K, Khan H, Atassi F, Kwak C, Jankovic J. Daytime sleepiness and other sleep disorders in Parkinson's disease. Neurology. 2001 Oct 23;57(8):1392-6. doi: 10.1212/wnl.57.8.1392. PMID 11673578
- [Background] King AC, Oman RF, Brassington GS, Bliwise DL, Haskell WL. Moderate-intensity exercise and self-rated quality of sleep in older adults. A randomized controlled trial. JAMA. 1997 Jan 1;277(1):32-7. PMID 8980207
- [Background] Li F, Fisher KJ, Harmer P, Irbe D, Tearse RG, Weimer C. Tai chi and self-rated quality of sleep and daytime sleepiness in older adults: a randomized controlled trial. J Am Geriatr Soc. 2004 Jun;52(6):892-900. doi: 10.1111/j.1532-5415.2004.52255.x. PMID 15161452
- [Background] Reid KJ, Baron KG, Lu B, Naylor E, Wolfe L, Zee PC. Aerobic exercise improves self-reported sleep and quality of life in older adults with insomnia. Sleep Med. 2010 Oct;11(9):934-40. doi: 10.1016/j.sleep.2010.04.014. Epub 2010 Sep 1. PMID 20813580
- [Background] Baatile J, Langbein WE, Weaver F, Maloney C, Jost MB. Effect of exercise on perceived quality of life of individuals with Parkinson's disease. J Rehabil Res Dev. 2000 Sep-Oct;37(5):529-34. PMID 11322151
- [Background] Rodrigues de Paula F, Teixeira-Salmela LF, Coelho de Morais Faria CD, Rocha de Brito P, Cardoso F. Impact of an exercise program on physical, emotional, and social aspects of quality of life of individuals with Parkinson's disease. Mov Disord. 2006 Aug;21(8):1073-7. doi: 10.1002/mds.20763. PMID 16637049